CLINICAL TRIAL: NCT06249763
Title: Effects of Dietary Gluten on Gastrointestinal Symptoms in Ulcerative Colitis: a Randomised Crossover Trial.
Brief Title: Effects of Gluten Free Diet in Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Colitis-Crohn Foreningen (Other); Hospital of Southern Jutland (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Vibeke Andersen, Professor, University of Southern Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Gluten-UC
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis
Keywords: Biomarkers; Treatment outcome; Gluten; Diet; Microbiome; Gastrointestinal symptoms; Fatigue
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Fatigue | interventions — Glutens; Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are randomised by an external source. Participants, care provider, investigator and outcomes assessor will be blinded to the randomisation. In case of adverse events, the randomization will be revealed to the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High gluten (Experimental): Participants complete both study arms in a crossover design separated by a washout period.
  Interventions: Dietary Supplement: Gluten free diet
- Gluten free (Placebo Comparator): Participants complete both study arms in a crossover design separated by a washout period.
  Interventions: Dietary Supplement: High gluten diet

INTERVENTIONS:
Dietary Supplement: High gluten diet — Trial period A: gluten free diet added daily granola bars with 10 g gluten/day (intervention).
  Other Names: G (gluten)
  Arms: Gluten free
Dietary Supplement: Gluten free diet — Trial period B: gluten free diet added daily granola bars with <1 g gluten/day (placebo).
  Other Names: GF (gluten free)
  Arms: High gluten

SUMMARY:
The goal is to evaluate gastrointestinal symptoms and fatigue levels during a period of eating gluten free compared to a period of high gluten consumption in individuals with confirmed Ulcerative Colitis, and to identify clinical characteristics in the blood and microbiome of those improving from a gluten free diet. The main questions, the project aims to answer are:

* What is the effect of eating gluten free on patient-reported gastrointestinal symptoms in patients with Ulcerative Colitis?
* What is the effect of eating gluten free on patient-reported fatigue levels in patients with Ulcerative Colitis?
* What are clinical differences between those improving and not improving on fatigue levels and gastrointestinal symptoms?

During two study periods of one week each, participants will be eating gluten free supplemented with daily granola bars without and with high gluten content, respectively. During each active week, participants are asked to:

* Eat gluten free and two daily granola bars delivered by the research team
* Collect blood, stool and urine samples
* Answer questionnaires about their symptoms, disease course, habitual lifestyle, and compliance to the protocol

DETAILED DESCRIPTION:
Introduction: To meet the growing demand for lifestyle recommendations among patients Ulcerative Colitis (UC) for managing their symptoms and wellbeing, this study aims to evaluate the use of the gluten free diet in the management of UC. Exposure to gluten can activate pro-inflammatory signals in the epithelium that induce mucosal damage, and the protein has previously been associated with disease activity in inflammatory bowel disease, including UC. A suggested pathway for the interaction between disease course and gluten intake is via mucosal damage followed by a flow of pathogens across the intestinal barrier.

To our knowledge, the effect of gluten on UC disease course is not fully understood, and clinical characteristics of patients benefitting from the gluten free diet has not yet been studied. To the patients, fatigue and pain from the gastrointestinal tract are the most burdensome symptoms of UC affecting life quality and restricting everyday activities for the patients. Hence, this study aims to evaluate the effects of dietary gluten in the management of gastrointestinal symptoms and fatigue in UC, and to identify clinical characteristics of patients with UC benefitting from eating gluten free.

Design: In this crossover randomized trial, the outcomes will be assessed after a one-week period of a high-gluten diet and a one-week period of a gluten free diet. Participants and study personnel will be blinded to the dietary intake by granola bars supplementing a complete gluten free diet. The intake of dietary fibres and fructans will be controlled and monitored and controlled for.

Setting: Participants will be recruited from the outpatient clinics for Gastrointestinal Diseases at Hospital Sønderjylland (Hospital of Southern Jutland) in the city of Aabenraa from from January to May 2024. Data collection will be completed in 2024.

Clinical data consist of personal data, patient-reported data on disease activity, gastrointestinal symptoms, fatigue level, health related quality of life and dietary intake, biomarkers in blood, urine and faeces, and protocol compliance measures. Information registered by clinicians and technicians will be transferred from paper format to electronic format using either double entry of data or automated forms processing.

Biologic material consist of blood, faeces and urine samples. All data are treated confidentially and stored according to the Danish Data Protection Regulation and Data Protection Law.

Sample size considerations: The sample size was based on a mixed effect model, hence we used Monte Carlo simulation to estimate the sample size. We defined a clinical significant improvement on the GSRS as a difference between groups of 1.0 in the mean score with an assumed standard deviation of 1.8 units and an interclass correlation of 0.56. Under these assumptions 15 participants were estimated to achieve a power of 80% at a 5%-significance level with a two-sided p-value based on a likelihood ratio test. However, if the correlation between the measures are 0.75 (instead of 0.50), 15 participants would likely respond to a statistical power of 99%.

Project organization: The project is part of a PhD (doctor of philosophy) study. Collaborators are specialists from the gastrointestinal, biochemical and microbiology departments involved in the project and professors in biostatistics and food sciences.

The study is approved by the local Ethics Committee (S-20210174) and the local Data Agency (22/39335). The study findings will be disseminated in peer-reviewed journals, via patient associations, and presented at national and international conferences.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Ulcerative Colitis (UC)
* Language: Can read and understand Danish
* Treatment: No intention to change dose of, begin, or switch medication and biologic treatment within one month after inclusion
* Treatment: Medical and/or biologic treatment type and dose stable for at least 8-16 weeks prior to inclusion depending on the type of treatment

Exclusion Criteria:

* Age: <18 years
* Severe disease activity defined by 6 or more bloody stools per day and/or night and one of the following: fever, pulse ≥ 90, C-reactive protein (CRP) ≥ 30mg/L by the time of inclusion
* Treatment: Have received antibiotic treatment within 4 weeks prior to inclusion
* Treatment: Previous operation for UC
* Concomitant diagnoses: Coeliac Disease (positive Immunoglobolin A against transglutaminase, TGA-IgA) or any cancer diagnosis
* Other: Taking probiotics, are pregnant or breastfeeding, or have nut or wheat allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | 1 week
  The Gastrointestinal Symptom Rating Scale (GSRS)

SECONDARY OUTCOMES:
Fatigue | 1 week
  Section I of the Inflammatory Bowel Disease Fatigue patient self-assessment scale (IBD-F) modified to assess the previous week
Disease activity | 1 week
  Simple Clinical Colitis Activity Index (SCCAI)
Symptom burden | 1 week
  Symptom burden measured on the Short Health Scale (SHS)
Functional status | 1 week
  Functional status measured on the Short Health Scale (SHS)
Disease-related health burden | 1 week
  Disease-related health burden measured on the Short Health Scale (SHS)
General well-being | 1 week
  General well-being measured on the Short Health Scale (SHS)
Joint pain | 1 week
  100 mm visual analogue scale (VAS)
Stool consistency | 1 week
  the Bristol Stool Form Scale (BSFS)
Faecal Calprotectin (f-Cal) | 1 week
  Intestinal inflammatory biomarker
C-reactive protein (CRP) | 1 week
  Acute phase reactant
Serum-Zonulin | 1 week
  Exploratory measure of intestinal permeability: Zonulin levels in blood and faeces
Faecal-Zonulin | 1 week
  Exploratory measure of intestinal permeability: Zonulin levels in blood and faeces
Dietary compliance: diet intake | 1 week
  Participant reported compliance to the diet (y/n), e.g. dietary gluten and fructan intake and the number of remaining granola bars by the end of a trial period
Urine-Gluten Immunogenic Peptides (GIP) | 1 week
  Supplementing dietary compliance measure: Presence of GIP in urine

OTHER OUTCOMES:
Microbiome data | 1 week
  Microbiome sequencing of urine and faecal samples
Potential biomarkers | 1 week
  Potential biomarkers in biologic material

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Andersen, Prof, Principal Investigator — University of Southern Denmark
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark, Denmark

DOCUMENTS (1):
  • Informed Consent Form (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT06249763/ICF_000.pdf